CLINICAL TRIAL: NCT04214379
Title: Evaluation of Polytetrafluoroethylene (Ptose-up) in Management of Severe Congenital Blepharoptosis
Brief Title: Management of Severe Congenital Blepharoptosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Farag Khalil Ibrahiem, Assistant Professor, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Oculoplastic Unit
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Blepharoptosis
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- severe congenital ptosis (Other): Patients with severe congenital ptosis with poor levator muscle function
  Interventions: Procedure: Ptosis surgery

INTERVENTIONS:
Procedure: Ptosis surgery — Frontalis sling surgery using pose-up and Wright's fascia-lata needle

SUMMARY:
Frontalis sling surgery was carried out using Ptose-up under general anaesthesia for patients with severe congenital ptosis.

DETAILED DESCRIPTION:
Frontalis sling surgery was carried out using Ptose-up for patients with severe congenital ptosis in 23 eyes of 15 patients and they followed up for at least 6 months to detect the success rate and if there is any postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Severe congenital blepharoptosis
* Poor levator muscle function
* No previous ptosis surgery

Exclusion Criteria:

* Patients with Jaw winking phenomenon
* Blepharophimosis syndrome
* Congenital myasthenia

Ages: 11 Months to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Improvement of ptosis | 3 months
  The average marginal reflex distance was improved from -0.8 mm preoperative to +2.73 mm after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Ibrahiem, MD, Principal Investigator — Minia University
Locations (1):
- Faculty of Medicine, Minya, Minya Governorate, Egypt